CLINICAL TRIAL: NCT05419622
Title: Analysis of Bronchial Remodeling Using Resonance Magnetic Imaging in Severe Asthmatic childrEn
Acronym: ARISE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2020/48
Record Dates: First submitted 2022-05-11; First posted 2022-06-15 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Asthma in Children
Keywords: asthma; children; serious; magnetic resonance imaging
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: Early study to evaluate the diagnostic and diagnostic performances of an imaging sequence, non-randomized, observational, prospective and bicentric.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- lung MRI (Experimental): The procedure under study is lung MRI, performed on a 1.5T magnet (AERA dot 1.5T, Siemens), without anesthesia and without injection or inhalation of contrast agent.
  Interventions: Biological: bronchial biopsies

INTERVENTIONS:
Biological: bronchial biopsies — This fibroscopy will make it possible to perform 4 bronchial biopsies at the level of the 4th bronchial generation (subsegmental bronchi), using suitable pediatric forceps.

SUMMARY:
This study is a diagnostic imaging pilot study evaluating performance of 3D-Ultrashort Time Echo (3D-UTE) Magnetic Resonance Imaging (MRI) for the diagnosis of bronchial remodeling in children with severe asthma. The primary objective is to compare bronchial parameters measured by 3D-UTE MRI according to the presence or the absence of bronchial remodeling determined on bronchial biopsies using immunohistochemistry, in severe asthmatic children.

DETAILED DESCRIPTION:
Background: Asthma is the most frequent chronic disease in childhood. Severe asthma accounts for only 5% of patients but more than half of the costs of the disease. It is characterized by bronchial remodeling, including an increase in bronchial smooth muscle (BSM) mass associated with an increase in bronchial smooth muscle cell proliferation. This increased cell proliferation has been related with an abnormal calcium homeostasis and an enhanced mitochondrial biogenesis. Moreover, the release of growth factors by inflammatory cells and bronchial epithelial cells reinforces BSM cell proliferation. BSM remodeling is correlated with the severity and poor control of the disease. In children, bronchial remodeling could be assessed by performing endobronchial biopsies during bronchoscopy. However, this method is invasive and cannot be repeated to follow the remodeling. Non-invasive quantification of proximal bronchial thickness by computed tomography (CT) has been demonstrated. However, CT was unable to differentiate bronchial inflammation from remodeling on the one hand, and, on the other hand, CT is a radiating examination, and the repetition of X-ray exposures can be a source of cancer. Recently, the team evaluated at the university hospital of Bordeaux new MRI sequences to obtain 3D high-resolution images (3D-UTE), close to that of CT. This 3D-UTE has the advantage of being performed without any injection or inhalation of contrast medium and non-irradiating. Moreover, MRI provides additional data on signal intensity or bronchial inflammation that is not accessible on CT imaging. However, to the best of our knowledge, the use of 3D -UTE high resolution MRI has not been demonstrated in a pediatric population with severe asthma.

Purpose: To compare bronchial parameters measured in 3D-UTE MRI according to the presence or not of bronchial remodeling measured by immunohistochemistry on bronchial biopsies obtained from severe asthmatic children.

Methods: The investigator's team therefore wishes to carry out pulmonary MRI without anesthesia, nor injection nor inhalation of contrast product in severe asthmatic children. Two sequences in axial cuts will be performed for a total duration of 12 minutes (6 minutes by sequence). Bronchial quantitative data obtained by MRI will be compared to those obtained from immunohistochemical analysis of bronchial biopsies performed during bronchoscopy. Severe asthmatic children requiring bronchoscopy will be identified during consultation or hospitalization relative of the disease. The inclusion visit (V1) will be performed during a consultation for asthma of the usual care of the child. Then, the second visit (V2) will correspond to the anesthesia consultation of the usual care of the child to check the absence of contraindications to anesthesia and bronchoscopy. The third visit (V3) will correspond to the pulmonary MRI and flexible bronchoscopy. According to the classic procedure, bronchoscopy will be performed during a hospitalization. The pulmonary MRI, as well as blood tests and lung function testing, will be performed at the beginning of the hospitalization, the day before the bronchoscopy. Children will be monitored 24 hours in hospitalization after the bronchoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Child from 6 to 17 years old
* Having informed consent signed by the holders of parental authority.
* Having a diagnosis of severe asthma according to the Global Initiative for Asthma (GINA) 2020;

  * Asthma: chronic inflammatory disease of the airways, defined mainly by respiratory symptoms such as wheezing, dyspnea, chest tightness and / or cough, which may vary in time and intensity associated with a limitation also varying in the time of expiratory flow.
  * Severe asthma: asthma which requires treatment with inhaled corticosteroids in high doses plus a second long-acting bronchodilator type controller, to maintain control of symptoms and / or whose control worsens if this treatment is reduced and / or which remains uncontrolled despite this treatment.
* Having to carry out as part of the current care a functional respiratory exploration;
* Should require as part of the routine care of a bronchial fibroscopy.

Exclusion Criteria:

* Patient without affiliation or not benefiting from a social security scheme;
* Patient being in a period of relative exclusion from another protocol;
* Patient born before 36 weeks of amenorrhea;
* Patient with a documented history of pulmonary fibrosis, primary pulmonary arterial hypertension, cystic fibrosis, pulmonary malformation or chronic viral infections (hepatitis, HIV);
* Patient presenting with an exacerbation of asthma requiring systemic corticosteroids within the previous 4 weeks;
* Patient with any dental, nasopharyngeal or bronchial infection with fever (> 39 ° C) requiring systemic antibiotics within the previous 4 weeks
* Patient with a contraindication to MRI:

  * Abdominal perimeter greater than 200 cm;
  * Claustrophobia or inability to lie still for 12 minutes;
  * Have a pacemaker or implantable defibrillator, intraocular metallic foreign body, intracranial metal clip, a pre-6000 Starr-Edwards type heart valve prosthesis, or a biomedical device such as an insulin pump or neurostimulator, cochlear implant and metal patch.
* Patient with a contraindication to anesthesia;
* Patient with a contraindication to bronchial fibroscopy following:

  * Abnormal hemostasis assessment;
  * Subject with cardiac pathology.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2023-06-08 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Measure of Bronchial thickness (BT) in UTE-T1 (in mm) | Day 30
  Mean (or median if the distribution is not normal) of the following candidate parameters measured on the 3D-UTE MRI performed either on the average of the 4th bronchial generation or on the only biopsied bronchus obtained at Visit 3:
  - Bronchial thickness (BT) in UTE-T1 (mm)
Measure of Signal strength of the bronchial wall (SB) in UTE-T1 (in milliseconds) | Day 30
  Mean (or median if the distribution is not normal) of the following candidate parameters measured on the 3D-UTE MRI performed either on the average of the 4th bronchial generation or on the only biopsied bronchus obtained at Visit 3:
  - Signal intensity of bronchial edema (SE) in T2- Turbo Spin-Echo (TSE) (second)
Measure of Volume of bronchial edema (VO) in T2-Turbo Spin-Echo (TSE) (in cubic millimeters) | Day 30
  Mean (or median if the distribution is not normal) of the following candidate parameters measured on the 3D-UTE MRI performed either on the average of the 4th bronchial generation or on the only biopsied bronchus obtained at Visit 3:
  - Volume of bronchial edema (VE) in T2-Turbo Spin-Echo (TSE) (mm^3)
Measure of Bronchial edema (SO) signal intensity in T2-Turbo Spin-Echo (TSE) (in milliseconds) | Day 30
  Mean (or median if the distribution is not normal) of the following candidate parameters measured on the 3D-UTE MRI performed either on the average of the 4th bronchial generation or on the only biopsied bronchus obtained at Visit 3:
  - Signal intensity of bronchial edema (SE) in T2-Turbo Spin-Echo (TSE) (second)

SECONDARY OUTCOMES:
Comparison each measurable values between 2 Physicians evaluated in the principal outcome measures | Day 30
  Intra-and inter-observer intraclass correlation coefficients of each of the parameters measured in 3D-UTE MRI, with their 95% confidence interval, and graphic representation of Bland and Altman
Measure of expiratory forced vital capacity (FVC) | Day 30
  Functional respiratory data
Measure of forced expiratory volume in one second (FEV1) | Day 30
  Functional respiratory data
Measure length of reticular basement membrane (RBM) completely denuded or covered by a single layer of basal cells with no intact ciliated or goblet cell over total basement membrane length | Day 30
  Values measured by immunohistochemistry to assess epithelial integrity in percent.
Measure of reticular basement membrane thickness (µm) | Day 30
  Values measured by immunohistochemistry
Measure of density of blood vessels (number/cm²) | Day 30
  Values measured by immunohistochemistry
Measure of normalized fibrosis area (%) | Day 30
  Values measured by immunohistochemistry
Measure of reticular basement membrane to bronchial smooth muscle distance (µm) | Day 30
  Values measured by immunohistochemistry

CONTACTS AND LOCATIONS:
Overall Officials: Fabien BEAUFILS, MD, Principal Investigator — University Hospital, Bordeaux
Locations (2):
- France (2):
  - CHU de Bordeaux - Explorations Fonctionnelles, Bordeaux
  - Centre Hospitalier de Saintonge, Saintes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bara I, Ozier A, Tunon de Lara JM, Marthan R, Berger P. Pathophysiology of bronchial smooth muscle remodelling in asthma. Eur Respir J. 2010 Nov;36(5):1174-84. doi: 10.1183/09031936.00019810. PMID 21037369
- [Result] Girodet PO, Ozier A, Bara I, Tunon de Lara JM, Marthan R, Berger P. Airway remodeling in asthma: new mechanisms and potential for pharmacological intervention. Pharmacol Ther. 2011 Jun;130(3):325-37. doi: 10.1016/j.pharmthera.2011.02.001. Epub 2011 Feb 17. PMID 21334378
- [Result] Bossley CJ, Fleming L, Gupta A, Regamey N, Frith J, Oates T, Tsartsali L, Lloyd CM, Bush A, Saglani S. Pediatric severe asthma is characterized by eosinophilia and remodeling without T(H)2 cytokines. J Allergy Clin Immunol. 2012 Apr;129(4):974-82.e13. doi: 10.1016/j.jaci.2012.01.059. Epub 2012 Mar 3. PMID 22385633
- [Result] Benlala I, Dournes G, Girodet PO, Benkert T, Laurent F, Berger P. Evaluation of bronchial wall thickness in asthma using magnetic resonance imaging. Eur Respir J. 2021 Dec 31;59(1):2100329. doi: 10.1183/13993003.00329-2021. Print 2022 Jan. No abstract available. PMID 34049945
- [Result] Dournes G, Yazbek J, Benhassen W, Benlala I, Blanchard E, Truchetet ME, Macey J, Berger P, Laurent F. 3D ultrashort echo time MRI of the lung using stack-of-spirals and spherical k-Space coverages: Evaluation in healthy volunteers and parenchymal diseases. J Magn Reson Imaging. 2018 Dec;48(6):1489-1497. doi: 10.1002/jmri.26212. Epub 2018 Sep 11. PMID 30203889